CLINICAL TRIAL: NCT01968187
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Effectiveness of Intranasal Carbetocin in Subjects With Prader-Willi Syndrome (PWS)
Brief Title: Treatment of Hyperphagia Behavioral Symptoms in Children and Adults Diagnosed With Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000114
Record Dates: First submitted 2013-10-09; First posted 2013-10-23 (Estimated); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hyperphagia in Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Carbetocin (FE 992097) (Experimental)
  Interventions: Drug: FE 992097
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FE 992097 — Each spray pump actuation delivered a 50 μL volume of solution that contained 1.6 mg carbetocin (FE 992097); each dose consisted of 3 spray pump actuations in each nostril that delivered a total of 9.6 mg carbetocin.
  Parents were instructed to administer 3 intranasal spray actuations in each nostril 3 times daily before meals for 14 days.
  Arms: Carbetocin (FE 992097)
Drug: Placebo — Each spray pump actuation delivered a 50 μL volume of sterile sodium chloride solution 0.9%; each dose consisted of 3 spray pump actuations in each nostril.
  Parents were instructed to administer 3 intranasal spray actuations in each nostril 3 times daily before meals for 14 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of intranasal FE 992097 in children and adults with Prader-Willi Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 10-18 years of age (both inclusive)
* Genetically confirmed diagnosis of Prader-Willi Syndrome
* Determined to be in nutritional phase 3 Prader-Willi Syndrome based on Miller et al, 2011

Exclusion Criteria:

* Known genetic, hormonal, or chromosomal cause of cognitive impairment other than Prader-Willi Syndrome
* Presence of currently active psychotic symptoms
* Presence of any cardiovascular disorders, epilepsy, frequent migraines or severe asthma
* Previous diagnosis of autism spectrum disorder by a qualified healthcare provider
* Prior or concomitant use of a selective serotonin reuptake inhibitor (SSRI) or selective norepinephrine reuptake inhibitor (SNRI), antipsychotic medication, wakefulness-promoting drug, or thyroid hormone unless dosage has been stable ≥6 months at time of screening

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2014-07-16 (Actual); Study Completion 2014-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (3):
- United States (3):
  - Florida University, Gainesville, Florida
  - Winthrop University, Mineola, New York
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dykens EM, Miller J, Angulo M, Roof E, Reidy M, Hatoum HT, Willey R, Bolton G, Korner P. Intranasal carbetocin reduces hyperphagia in individuals with Prader-Willi syndrome. JCI Insight. 2018 Jun 21;3(12):e98333. doi: 10.1172/jci.insight.98333. eCollection 2018 Jun 21. PMID 29925684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in the United States, and a total of 3 sites randomized subjects to the trial between Jan 2014 to Jul 2014.
Pre-assignment Details: In total, 38 subjects were screened and randomized. One subject in the Carbetocin (FE 992097) arm was randomized in error and did not receive the investigational medicinal product (IMP), and was listed as a screening failure. Of the randomized subjects, 37 subjects were exposed to IMP: 17 to Carbetocin (FE 992097) and 20 to placebo.
Groups:
- Carbetocin (FE 992097): Each spray pump actuation delivered a 50 μL volume of solution containing 1.6 mg carbetocin (FE 992097); each dose consisted of 3 spray pump actuations in each nostril delivering a total of 9.6 mg carbetocin.
  Parents were instructed to administer 3 intranasal spray actuations in each nostril 3 times daily before meals for 14 days.
Period: Overall Study
Arm/Group | Carbetocin (FE 992097) | Placebo
Started | 18 | 20
Treated (A total of 18 subjects were randomized. However, 1 was randomized in error and not treated.) | 17 | 20
Completed | 17 | 19
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population included the safety analysis set (SAS) which consisted of all subjects who received any amount of the IMP. Analyses for the safety population were conducted according to the actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbetocin (FE 992097) | Placebo | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (2.45) | 13.6 (2.52) | 13.7 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.72 (5.947) | 25.66 (7.537) | 25.69 (6.760)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hyperphagia in Prader-Willi Syndrome (PWS) Questionnaires- Responsiveness (HPWSQ-R) Total Score at End-of-treatment (Day 15)
Description: The HPWSQ-R is an 11-item questionnaire examining the psychological, developmental, and neurobiological correlates of hyperphagia in PWS. The items are classified into 3 domains; behavior, drive, and severity with each item rated on a five-point scale (1: not at all/none of the time/extremely easy to 5: extremely/all of the time/extremely hard). The questionnaire was completed by the parent/caregiver using a 1-week recall period. Total score was the sum of all the items in the three domains and ranged from 11 (no hyperphagia behaviors) to 55 (most severe hyperphagia behaviors).
  Change from baseline in HPWSQ-R Total Score at Day 15 is presented for this outcome measure.
Time Frame: From Day 1 (baseline) to Day 15
Population: The analysis population included the full analysis set (FAS) which consisted of all subjects in the safety population who had the primary efficacy endpoint measured (at baseline and phone call [Day 8] ±1 or Day 15). Analyses for the FAS were conducted according to the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Carbetocin (FE 992097) | Placebo
Number analyzed (Participants) | 17 | 20
score on a scale | -15.6 (3.06) | -8.9 (2.61)
Statistical Analysis 1: Comparison: Carbetocin (FE 992097) vs Placebo; Test type: Other; p = 0.0290, ANCOVA; Treatment groups were compared using ANCOVA model with treatment and site as fixed effect and HPWSQ-R total score at baseline as covariate; LS Mean Difference = -6.7, 90% CI 1-sided [upper limit -2.2]

2. Secondary Outcome: Clinical Global Impression- Improvement After Treatment (CGI-I) Score at End-of-treatment (Day 15)
Description: The Clinical Global Impression (CGI) scale consists of a 7-point clinician rating of illness severity (1 = normal, not at all ill, 7 = among the most extremely ill patients), at the beginning of the trial (baseline) - Clinical Global Impression-Severity Rating (CGI-S) and a 7-point clinician rating of improvement of patient condition (1=very much improved since baseline/initiation of treatment, 7=very much worse from baseline), during and at the end of the trial (Day 15) - CGI-I.
  The CGI-I score at Day 15 is presented for this outcome measure.
Time Frame: At Day 15
Population: The analysis population included the full analysis set (FAS) which consisted of all subjects in the safety population who had the primary efficacy endpoint measured (at baseline and phone call [Day 8] ±1 or Day 15). Analyses for the FAS were conducted according to the randomized treatment.
  Number of subjects analyzed signifies those subjects who were evaluable for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Carbetocin (FE 992097) | Placebo
Number analyzed (Participants) | 16 | 19
score on a scale | 2.7 (0.49) | 3.6 (0.43)
Statistical Analysis 1: Comparison: Carbetocin (FE 992097) vs Placebo; Test type: Other; p = 0.0233, ANCOVA; Treatment groups were compared using ANCOVA model with treatment and site as fixed effects and CGI-S score as a covariate; LS Mean Difference = -0.8, 90% CI 1-sided [upper limit -0.3]

3. Secondary Outcome: Change From Baseline in HPWSQ-R Domain Scores (Behavior, Drive and Severity) at End-of-treatment (Day 15)
Description: The HPWSQ-R is an 11-item questionnaire examining the psychological, developmental, and neurobiological correlates of hyperphagia in PWS. The items were classified into 3 domains; behavior, drive, and severity with each item rated on a five-point score range from 1 (not at all/none of the time/extremely easy) to 5 (extremely/all of the time/extremely hard). The questionnaire was completed by the parent/caregiver using a 1-week recall period.
  Changes in the HPWSQ-R Total Score and in the Domain Scores (behavior, drive, and severity) at Day 15 is presented for this outcome measure.
  HPWSQ-R Behavior, Drive and Severity scores range from 5-25, 4-20, and 2-10, respectively, with higher scores indicating a worse outcome.
  Change from baseline is presented = (Day 15 score minus Baseline score).
Time Frame: From Day 1 (baseline) to Day 15
Population: The analysis population included the FAS which consisted of all subjects in the safety population who had the primary efficacy endpoint measured (at baseline and phone call [Day 8] ±1 or Day 15). Analyses for the FAS were conducted according to the randomized treatment.
Measure: Least Squares Mean (Full Range); unit: score on a scale
Arm/Group | Carbetocin (FE 992097) | Placebo
Number analyzed (Participants) | 17 | 20
score on a scale
  Behavior | -5.9 [-16 to 3] | -3.9 [-14 to 3]
  Drive | -4.5 [-13 to 3] | -2.9 [-16 to 3]
  Severity | -3.3 [-7 to 2] | -1.8 [-7 to 3]
Statistical Analysis 1: Comparison: Carbetocin (FE 992097) vs Placebo; HPWSQ-R Domain score: Behavior; Test type: Other; p = 0.1172, ANCOVA; Treatment groups were compared using ANCOVA model with treatment and site as fixed effects and HPWSQ-R domain score at baseline as a covariate; LS Mean Difference = -2.0, 90% CI 1-sided [upper limit 0.2]
Statistical Analysis 2: Comparison: Carbetocin (FE 992097) vs Placebo; HPWSQ-R Domain score: Drive; Test type: Other; p = 0.1436, ANCOVA; Treatment groups were compared using ANCOVA model with treatment and site as fixed effects and HPWSQ-R domain score -at baseline as a covariate; LS Mean Difference = -1.6, 90% CI 1-sided [upper limit 0.3]
Statistical Analysis 3: Comparison: Carbetocin (FE 992097) vs Placebo; HPWSQ-R Domain score: Severity; Test type: Other; p = 0.0248, ANCOVA; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = -1.5, 90% CI 1-sided [upper limit -0.5]

4. Secondary Outcome: Change From Baseline in Children's Yale-Brown Obsessive Compulsive Scale Score (CY-BOCS) at End-of-treatment (Day 15)
Description: The CY-BOCS is a clinician rated, semi-structured inventory of specific symptoms and symptom severity in pediatric obsessive-compulsive disorder (OCD). Total scores on the CY-BOCS are calculated using a symptom checklist and severity scale. The 10 severity items are summed to produce an Obsessions Severity Score (5 items), Compulsions Severity Score (5 items), and Total score (sum of all 10 severity items).
  The total score is calculated by summing the 10 individual scores and ranges from 0 (no obsessions or compulsions) to 40 (most severe OC).
Time Frame: From Day 1 (baseline) to Day 15
Population: The analysis population included the FAS which consisted of all subjects in the safety population who had the primary efficacy endpoint measured (at baseline and phone call [Day 8] ±1 or Day 15). Analyses for the FAS were conducted according to the randomized treatment.
  Number of subjects analyzed signifies those subjects who were evaluable for this endpoint
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Carbetocin (FE 992097) | Placebo
Number analyzed (Participants) | 16 | 19
score on a scale | -8.8 (2.29) | -2.6 (1.82)
Statistical Analysis 1: Comparison: Carbetocin (FE 992097) vs Placebo; Test type: Other; p = 0.0047, ANCOVA; From ANCOVA model with treatment and site as fixed effects and CY-BOCS total score at baseline as a covariate; LS mean difference = -6.2, 90% CI 1-sided [upper limit -3.3]

5. Secondary Outcome: Change From Baseline in the Food Domain Score of the Reiss Profile at End-of-treatment (Day 15)
Description: The Food Domain Score of the Reiss Profile consisted of 7 questions that pertain to food seeking behavior. The questions were rated on a five point scale ranging from -2 (strongly disagree; this phrase is not at all characteristic of the person) to 2 (strongly agree; this phrase is definitely characteristic of the person). Total score was defined as the sum of all individual item scores. The total score ranged from -14 to 14 with higher scores indicating higher severity.
  Change from baseline in Food Domain of the Reiss Profile at Day 15 is presented for this outcome measure.
Time Frame: From Day 1 (baseline) to Day 15
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Carbetocin (FE 992097) | Placebo
Number analyzed (Participants) | 16 | 19
score on a scale | -6.9 (1.94) | -2.5 (1.55)
Statistical Analysis 1: Comparison: Carbetocin (FE 992097) vs Placebo; Test type: Other; p = 0.0132, ANCOVA; Compared using ANCOVA model with treatment and site as fixed effects and Food Domain Score of Reiss Profile at baseline as a covariate; LS mean difference = -4.4, 90% CI 1-sided [upper limit -1.9]

ADVERSE EVENTS:
Time Frame: The adverse events (AEs) were recorded from signing of the informed consent until the Day 19 follow-up phone call.
Description: Adverse events that began during the Treatment Period (period during which a subject received IMP) or worsening of a pre-existing medical condition (treatment-emergent AEs) are presented for the SAS.
Arm/Group | Carbetocin (FE 992097) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 7/17 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbetocin (FE 992097) (N=17) | Placebo (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (8) | 6 (18)
Dysgeusia (Nervous system disorders) | 1 (9) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT01968187/Prot_SAP_000.pdf